CLINICAL TRIAL: NCT02149563
Title: Oxygen Therapy in Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2014-04-07; First posted 2014-05-29 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Depression, Normobaric Hyperoxia.
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): One hundred participants will receive home treatment with oxygen-enriched air (40% O2) through a nasal tube during the night (7 hours) for one month.
  Interventions: Device: oxygen-enriched air -Normobaric hyperoxia treatment for depression
- Placebo (Placebo Comparator): 100 participants will receive regular air treatment (21% O2) through a nasal tube (identical to the procedure providing 40% O2) for one month
  Interventions: Device: oxygen-enriched air -Normobaric hyperoxia treatment for depression

INTERVENTIONS:
Device: oxygen-enriched air -Normobaric hyperoxia treatment for depression — Forty percent oxygen or regular air will be supplied from oxygen concentrators, through standard plastic nasal prongs, at a flow rate of 5 liters/minute, for 7 hours a day, throughout the night.
  Other Names: Oxygen-enriched air provided by oxygen concentrators to improve symptoms of patients with depression.

SUMMARY:
The major objective of the present study is to examine the influence of normobaric hyperoxia treatment on the symptoms of patients diagnosed with depression members of Clalit Health Services. The investigators hypothesize that normobaric hyperoxia treatment will improve the symptoms of patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-65 years diagnosed with mild to moderate depression.

Exclusion Criteria:

* Patients with oxygen saturation below 95%;
* An unstable mental (psychiatric) condition
* A psychiatric condition that requires a change in pharmacotherapy (importantly - medications will not be changed in patients who will be enrolled to the study)
* Acute or chronic respiratory disease
* Any severe physical illness
* Suicidal thoughts or attempts
* Drug abuse
* Obesity (BMI over 30)
* Inability to cease smoking during night hours while participants are supposed to be using the oxygen/air supplementing machine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HRSD)-changes in patients' depression. | Baseline (time zero), 2 weeks and 4 weeks
  HRSD will be used to assess changes in patients' condition. Assessment will be performed at 3 time points: baseline (time zero), 2 weeks and 4 weeks after treatment initiation, by a trained psychiatric nurse blind to the patient's treatment status.

CONTACTS AND LOCATIONS:
Locations (1):
- Clalit Health Services in the Southern region, Beersheba, Israel

REFERENCES:
- [Derived] Bloch Y, Belmaker RH, Shvartzman P, Romem P, Bolotin A, Bersudsky Y, Azab AN. Normobaric oxygen treatment for mild-to-moderate depression: a randomized, double-blind, proof-of-concept trial. Sci Rep. 2021 Sep 23;11(1):18911. doi: 10.1038/s41598-021-98245-9. PMID 34556722